CLINICAL TRIAL: NCT02756533
Title: Impact of a Telemonitoring Program on the Rate of Hospitalizations for Worsening of Cardio-respiratory Symptoms in COPD Patients Treated at Home by Long-term Non-invasive Ventilation (NIV): a Randomized Controlled Trial
Brief Title: Impact of a Telemonitoring Program on the Rate of Hospitalizations for Worsening of Cardio-respiratory Symptoms in COPD Patients Treated at Home by Long-term Non-invasive Ventilation (NIV)
Acronym: EXA-VNI2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: pilot feasibility study completed
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Philips Healthcare (Industry); AGIR à Dom (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 38RC15.179
Record Dates: First submitted 2016-03-22; First posted 2016-04-29 (Estimated); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telemonitoring (Experimental): Telemonitoring of daily parameters recorded by NIV, transmitted to a remote monitoring platform. When an alert is received the patient is contacted by phone by a nurse to evaluate the worsening of symptoms. Information are transferred to a referent physician for further medical care if needed.
  Interventions: Other: Telemonitoring of daily parameters recorded by NIV
- control (Placebo Comparator): Telemonitoring of daily parameters by NIV, transmitted to a remote monitoring platform with no generation of alerts.
  Phone calls to patient during the follow-up like "false alerts" for the blind procedure.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Telemonitoring of daily parameters recorded by NIV — Daily telemonitoring of breathing rate, % of trigger cycles, daily usage of the NIV will go through an algorithm generating alerts when variations will go beyond normal. When an alert is received, a nurse will evaluate the symptoms of the patient by a standardized phone call questionnaire. The results will be transmitted to a referent practitioner who will decide what the patient should do.
  Recommendations will be transferred to the patient within 36 hours.
  Arms: Telemonitoring
Other: Placebo — Daily telemonitoring of breathing rate, % of trigger cycles, daily usage of the NIV will go through an algorithm generating alerts when variations will go beyond normal. Alerts will only be collected, the patient will not be contacted by phone during the alert.
  Arms: control

SUMMARY:
COPD is characterized by non-reversible chronic airway obstruction. Its evolution is punctuated by successive exacerbations precipitating the progression of the disease and its co-morbidities. The most severe exacerbations are the source of frequent hospitalizations that strongly affect the patient's quality of life and are associated with increased mortality. The diagnosis of exacerbation is mainly clinical but patients frequently consult their doctor too late which may lead to delays in care. However, the early detection and management of these exacerbations can reduce their impact and in particular avoid hospitalization or shorten their duration.

In France, long term Non-Invasive Ventilation (NIV) is a widely used treatment modality in COPD patients with chronic alveolar hypoventilation who have frequent exacerbations. The investigators have demonstrated in a previous study that the analysis of parameters from software embedded in the NIV device can reliably predict the occurrence of an exacerbation. The investigators hypothesize that the daily transmission via a telemonitoring platform of the ventilation parameters of patients, together with an ad hoc warning system, would reduce the rate of hospitalization for COPD patients treated at home with NIV thanks to the early detection and early treatment of these exacerbations.

The purpose of the study is to compare if a program of telemonitoring using the parameters stored by the NIV impact the rate of hospitalization for worsening of cardiorespiratory symptoms in COPD patients versus standard care over a one year period.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is characterized by non-reversible chronic airway obstruction associated with co-morbidities and is the third leading cause of death worldwide. Its evolution is punctuated by successive exacerbations precipitating the progression of the disease and its co-morbidities. The most severe exacerbations are the source of frequent hospitalizations that strongly affect the patient's quality of life and are associated with increased mortality. The diagnosis of exacerbation is mainly clinical but patients frequently consult their doctor too late which may lead to delays in care. However, the early detection and management of these exacerbations can reduce their impact and in particular avoid hospitalization or shorten their duration.

In France, long term Non-Invasive Ventilation (NIV) is a widely used treatment modality in COPD patients with chronic alveolar hypoventilation who have frequent exacerbations. In France, 7000-10000 COPD patients are currently treated with NIV. Recent NIV respirators are fitted with embedded software that provides details on treatment adherence (daily use, number of sessions/day, number of days of use over a given period etc) and on a number of ventilatory parameters measured during treatment (minute ventilation, tidal volume, respiratory rate, leaks, cycles triggered by the patient, etc.).

In a preliminary study, including more than 60 COPD patients treated with NIV, the investigators demonstrated that the analysis of parameters from software embedded in the NIV device can reliably predict the occurrence of an exacerbation in following five days.

The investigators hypothesize that the daily transmission via a telemonitoring platform of the ventilation parameters of patients, together with an ad hoc warning system, would reduce the rate of hospitalization for COPD patients treated at home with NIV thanks to the early detection and early treatment of these exacerbations.

The physiological and symptomatic changes that accompany an exacerbation can be detected by daily questionnaires, monitoring devices worn by the patient or easy to use appliances (respiratory rate sensor, touch pad for daily symptoms). These expensive devices require active patient involvement and a certain degree of skill by the patients, which limits their use. The main innovation of this project is that patients already have NIV treatment reimbursed by their health insurance and no further action will be required on the part of the patient to detect worsening. Changes recorded by the ventilator settings will trigger an alert and if needed early and appropriate patient care can be initiated.

Main objective:

The purpose of the study is to compare if a program of telemonitoring using the parameters stored by the NIV impact the rate of hospitalization for worsening of cardiorespiratory symptoms in COPD patients versus standard care over a one year period.

ELIGIBILITY:
Inclusion Criteria:

* COPD
* Treated by long term NIV
* Compliance over 0h
* Hospitalized for worsening of cardio-respiratory symptoms at least once during the past year
* With social security coverage

Non inclusion Criteria:

* Evolutionary pathology (excluding COPD) may be life-threatening in the short term (1 year) (cancer, neuromuscular disease rapidly changing) (doctor's discretion)
* Patients whom referring general practitioner or pulmonologist is refusing to participate
* Person deprived of liberty
* Major protected by law
* Pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2020-07-06 (Actual)

PRIMARY OUTCOMES:
Number of hospitalizations for worsening for cardio-respiratory symptoms. | one year
  An hospitalization being an entry in any hospital or clinic, whatever the length of the stay. The validation of cardiorespiratory worsening being the reason of the hospitalization will be done by a single independent retrospective committee of two doctors. The doctors won't be investigators of the study.Comparison between the two arms will be done.

SECONDARY OUTCOMES:
Number of un-programmed hospitalizations or death | one year
  Comparison between the two arms
External validation of the algorithm to early detect COPD exacerbation by all parameters recorded by NIV of both groups of patients | one year
  all parameters recorded by NIV done will be analyzed according to COPD exacerbations date validated by a single independent retrospective committee of two doctors. The predictive value and sensitivity and the specificity of individual parameters with different algorithm on the previous days of COPD exacerbation will be analyzed. Composite scores of several parameters will be analyzed.
Length of hospitalization for worsening of cardio-respiratory symptoms | one year
  Comparison between the two arms
medical cost | one year
  Comparison between the two arms
Quality of life assessed by SRI (Severe respiratory Insufficiency) score | 1 year
  Comparison between the two arms of the scores of the SRI questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis Pépin, Pr MD PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Grenoble University Hospital, Grenoble, France

IPD SHARING:
Plan to Share IPD: No